CLINICAL TRIAL: NCT04743999
Title: Prospective Evaluation of Quality of Life and Treatment-related Side Effects of Women Undergoing Multimodality Treatment for Advanced Stage Endometrial Carcinoma
Brief Title: Evaluation of Outcomes in Women Undergoing Multimodality Treatment for Advanced Stage Endometrial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Mohamed Elshaikh, Senior Staff Physician, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13551
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quality of life evaluation (Experimental): This prospective arm will consist of evaluating quality of life outcomes in women in women with advanced endometrial cancer undergoing adjuvant concurrent chemotherapy with carbo/Taxol and radiation therapy. Assessments will occur following surgery (baseline), 3, 6, 12, and 24 months.
  Interventions: Other: Quality of life questionnaire

INTERVENTIONS:
Other: Quality of life questionnaire — We will evaluate patients' quality of life with a series of questionnaires at baseline, 3, 6, 12, and 24 months after surgical staging. These are prospectively validated questionnaires and include FACT-G (physical and functional well-being sections), FACT-En (additional concerns section), FACT/GOG-NTX-4 (additional concerns section), and FACT-C (items C3 and C5).These sections will be combined into one single form for ease of completion for the patients (a total of 36 items).

SUMMARY:
Patients with FIGO stage III endometrial carcinoma often require multimodality adjuvant therapy to improve survival and recurrence rates; however, the optimal adjuvant therapy sequence is yet to be established.

Several studies have tried to answer this question including RTOG 9708, PORTEC-3, and GOG 258. Collectively, these studies show that concurrent chemotherapy and radiation (chemoRT) with cisplatin followed by additional chemotherapy (CT) and CT alone are acceptable regimens. However, both strategies show that distant recurrence remains a problem when CT is delayed after RT, and local control is compromised without RT.

We wish to prospectively assess outcomes of women with advanced endometrial carcinoma who receive concurrent chemoRT with a carboplatin/paclitaxel-based regimen.

A total of 60 patients with FIGO stage III uterine carcinoma will be prospectively enrolled after undergoing surgical staging (currently accruing). CT will start approximately 4 weeks after surgery. Patients will receive 6 cycles of carboplatin (AUC 6) and paclitaxel (175 mg/m2).

RT will be given during CT cycles 1-3. External beam RT will be given via intensity-modulated RT in once-daily fractions of 1.8-2.0 Gy for a total dose of 44-45 Gy to the pelvis (vaginal cuff, pelvic LN, and para-aortic lymph nodes). If there is grossly visible nodal disease seen at the time of treatment planning, a boost to 54 Gy will be given to those areas. If the patient has cervical stromal invasion, we will recommend that she receive a brachytherapy boost.

Data will be collected on OS and PFS endpoints. Data will also be collected on provider- and patient-reported treatment toxicity. Patients will receive a series of questionnaires at baseline, 3, 6, 12, and 24 months after surgery. These are prospectively-validated questionnaires and include FACT-G, FACT-En, FACT/GOG-NTX, and FACT-C.

For statistical analyses, continuous and categorical variables will be analyzed. Kaplan-Meier survival estimates will be calculated for local control and survival end points. For each patient, disease characteristics and adjuvant treatment will be placed in a simple logistic regression model for predicting survival endpoints. A multivariate analysis will be performed for exploratory purposes. Hazard ratios and 95% confidence intervals will be reported. Tests will be considered significant at p < 0.05.

DETAILED DESCRIPTION:
Purpose: To prospectively determine patients' quality of life (QOL) and treatment-related toxicity outcomes with adjuvant multimodality treatment (chemotherapy and radiation treatment) in women with advanced endometrial carcinoma after surgical staging.

Specific Aims:

1. To prospectively determine QOL after adjuvant treatment using the prospectively-validated FACT questionnaires at baseline, 3, 6, 12, and 24 months after surgical staging
2. To prospectively determine the rate of any grade 2 or higher treatment-related side effects: mainly bone marrow suppression, lymphedema, diarrhea, and others. Additionally, we will collect information about the rate of completion of planned adjuvant treatment (number of chemotherapy cycles, dose reduction or chemotherapy delay, radiation treatment interruption, etc.).
3. To prospectively collect survival outcome endpoints after adjuvant treatment (recurrence-free, disease-specific and overall survival).

Introduction and Rationale: Endometrial cancer is the most common gynecologic malignancy in the United States and ranks second in gynecologic cancer mortality following only ovarian cancer. More than 84% of patients present with International Federation of Gynecology and Obstetrics (FIGO) stage I-II disease. By definition, patients with advanced-stage uterine carcinoma (FIGO stages III-IV) are those with extrauterine disease and are at significant risk of dying from uterine cancer. They constitute a very heterogeneous group of patients with varying risk factors yielding highly variable clinical outcomes. Within the same FIGO stage, patients with disease involving multiple extrauterine sites fare worse compared to patients with involvement of a single site (1).

Postoperatively, patients with advanced stage disease often require adjuvant therapy(s) to reduce the chance of tumor recurrence with the potential to improve survival. However, the optimal adjuvant therapy is yet to be established with several options available for adjuvant treatment.

Rationale for multimodality treatment with chemotherapy and radiation treatment (CMT):

Current treatment recommendations for advanced stage endometrial cancer consist of multiple approaches including chemotherapy alone, radiotherapy (RT) alone, or combined modality treatment (CMT) (2).

GOG 122 study, which was a phase III trial, randomized patient with advanced endometrial carcinoma to adjuvant chemotherapy alone versus whole abdomen RT (WART). Outcomes of this study showed that the chemotherapy arm had an improved 5-year progression-free survival (PFS) and overall survival (OS) compared to RT alone. However, this trial showed that if chemotherapy is given alone, that rate of local recurrence approaches 20% (3).

The safety of CMT with concurrent chemotherapy and RT (chemoRT) was explored in RTOG 9708, which was a phase II trial that evaluated outcomes in patients receiving concurrent chemoRT. All patients received adjuvant pelvic RT (45 Gy) concurrent with cisplatin followed by four additional cycles of cisplatin and paclitaxel. The 4-year OS and PFS for patients with stage III disease were 77% and 72%, respectively. Rates of grade 1 toxicity were found in 16% of patients, grade 2 in 41%, grade 3 in 16%, and grade 4 in 5%. This study demonstrated that concurrent chemoRT is safe with excellent local control (4).

More recent studies have sought to compare chemoRT to chemotherapy or radiation alone. PORTEC-3 was a phase III randomized trial comparing adjuvant RT alone to concurrent chemoRT. The RT dose was 48.6 Gy in 27 fractions and chemotherapy was concurrent cisplatin followed by an additional 4 cycles of carboplatin and paclitaxel. For women with stage III disease, the addition of chemotherapy to radiation treatment showed benefit in terms of improvement in FFS. An analysis of toxicity outcomes found that 60% of patients in the chemoRT arm experienced a grade 3 or greater adverse event compared to 12% in the RT alone arm (p<0.0001) (5).

GOG 258 study was recently published and was similar to PORTEC-3 except that it compared concurrent chemoRT to adjuvant chemotherapy alone. Patients were randomized to receive concurrent chemoRT (45 Gy in 25 fractions concurrent with cisplatin followed by 4 cycles of carboplatin and paclitaxel) or chemotherapy alone. The results of this study showed that chemoRT was associated with a lower 5-year incidence of vaginal and regional lymphatic recurrence. However, distant recurrence rates were higher in the chemoRT arm compared to chemotherapy alone (6).

The above studies helped to establish concurrent chemoRT with cisplatin followed by adjuvant carboplatin/paclitaxel as a valid adjuvant treatment approach for women with advanced endometrial carcinoma.

A retrospective review from Washington University included 51 women with stage III-IV endometrial carcinoma who received CMT with carboplatin/paclitaxel-based regimen concurrent with RT and assessed survival and toxicity outcomes. The chemotherapy regimen given was carboplatin/paclitaxel for 4-6 cycles and RT was 48-51.2 Gy. Patients also received a vaginal brachytherapy boost. They found that 48 patients (94%) completed chemotherapy and 16 patients (30%) required chemotherapy dose-reduction. Thirty-four patients experienced grade 3-4 toxicities, most of which were hematologic. Over 80% of patients required leukocyte growth factor injections. There were seven late grade 3-4 toxicities (4 GI, 2 GU, and 1 ongoing neuropathy). They found a median PFS of 42.8 months, median OS of 44.9 months, and 3-year OS of 80% (7). This study suggests that concurrent chemoRT using a carbotaxol-based regimen has favorable outcomes, a tolerable side effect profile, and the potential to reduce overall treatment duration.

Building off of the results of the above retrospective study as well as the aforementioned randomized trials, we wish to prospectively assess outcomes of women with advanced endometrial carcinoma who receive the same concurrent chemoRT with a carboplatin/paclitaxel-based regimen.

ELIGIBILITY:
Inclusion Criteria:

* FIGO stage III uterine carcinoma
* candidates for combined modality treatment (surgery, chemotherapy with carbo/Taxol, and radiation therapy)

Exclusion Criteria:

* Patients who are not FIGO stage III
* patients with carcinosarcoma histology
* patients who are ineligible for combined modality treatment

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elshaikh, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elshaikh MA, Yashar CM, Wolfson AH, Cardenes HR, Erickson B, Jhingran A, Jolly S, Kidd E, Lee LJ, Mayr NA, Moore D, Rao GG, Small W Jr, Varia MA, Wahl AO, Yuh W, Gaffney DK; Expert Panel on Radiation Oncology-Gynecology:. ACR appropriateness Criteria(R) advanced stage endometrial cancer. Am J Clin Oncol. 2014 Aug;37(4):391-6. doi: 10.1097/COC.0000000000000098. PMID 24977691
- [Background] NCCN Guidelines Version 3.2019 Endometrial Carcinoma
- [Background] Randall ME, Filiaci VL, Muss H, Spirtos NM, Mannel RS, Fowler J, Thigpen JT, Benda JA; Gynecologic Oncology Group Study. Randomized phase III trial of whole-abdominal irradiation versus doxorubicin and cisplatin chemotherapy in advanced endometrial carcinoma: a Gynecologic Oncology Group Study. J Clin Oncol. 2006 Jan 1;24(1):36-44. doi: 10.1200/JCO.2004.00.7617. Epub 2005 Dec 5. PMID 16330675
- [Background] Greven K, Winter K, Underhill K, Fontenesci J, Cooper J, Burke T. Final analysis of RTOG 9708: adjuvant postoperative irradiation combined with cisplatin/paclitaxel chemotherapy following surgery for patients with high-risk endometrial cancer. Gynecol Oncol. 2006 Oct;103(1):155-9. doi: 10.1016/j.ygyno.2006.02.007. Epub 2006 Mar 20. PMID 16545437
- [Background] de Boer SM, Powell ME, Mileshkin L, Katsaros D, Bessette P, Haie-Meder C, Ottevanger PB, Ledermann JA, Khaw P, Colombo A, Fyles A, Baron MH, Jurgenliemk-Schulz IM, Kitchener HC, Nijman HW, Wilson G, Brooks S, Carinelli S, Provencher D, Hanzen C, Lutgens LCHW, Smit VTHBM, Singh N, Do V, D'Amico R, Nout RA, Feeney A, Verhoeven-Adema KW, Putter H, Creutzberg CL; PORTEC study group. Adjuvant chemoradiotherapy versus radiotherapy alone for women with high-risk endometrial cancer (PORTEC-3): final results of an international, open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2018 Mar;19(3):295-309. doi: 10.1016/S1470-2045(18)30079-2. Epub 2018 Feb 12. PMID 29449189
- [Background] Matei D, Filiaci V, Randall ME, Mutch D, Steinhoff MM, DiSilvestro PA, Moxley KM, Kim YM, Powell MA, O'Malley DM, Spirtos NM, Small W Jr, Tewari KS, Richards WE, Nakayama J, Matulonis UA, Huang HQ, Miller DS. Adjuvant Chemotherapy plus Radiation for Locally Advanced Endometrial Cancer. N Engl J Med. 2019 Jun 13;380(24):2317-2326. doi: 10.1056/NEJMoa1813181. PMID 31189035
- [Background] Wilkinson-Ryan I, Binder PS, Pourabolghasem S, Al-Hammadi N, Fuh K, Hagemann A, Thaker P, Schwarz J, Grigsby P, Mutch D, Powell M. Concomitant chemotherapy and radiation for the treatment of advanced-stage endometrial cancer. Gynecol Oncol. 2014 Jul;134(1):24-8. doi: 10.1016/j.ygyno.2014.05.002. Epub 2014 May 10. PMID 24823648

RESULTS

PARTICIPANT FLOW:
Period: Baseline Questionnaire
Arm/Group | Quality of Life Evaluation
Started | 9
Completed | 9
Not Completed | 0
Period: 3-month Questionnaire
Arm/Group | Quality of Life Evaluation
Started | 9
Completed | 8
Not Completed | 1
Not completed — Death | 1
Period: 6-month Questionnaire
Arm/Group | Quality of Life Evaluation
Started | 8
Completed | 7
Not Completed | 1
Not completed — Study terminated due to low accrual | 1
Period: 12-month Questionnaire
Arm/Group | Quality of Life Evaluation
Started | 7
Completed | 6
Not Completed | 1
Not completed — Study terminated due to low accrual | 1
Period: 24-month Questionnaire
Arm/Group | Quality of Life Evaluation
Started | 6
Completed | 1
Not Completed | 5
Not completed — Study terminated due to low accrual | 5

BASELINE CHARACTERISTICS:
Arm/Group | Quality of Life Evaluation
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Physical and Functional Well-being as Assessed by the FACT-G Questionnaire
Description: The Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire is a prospectively validated form that assesses physical side effects of treatment (eg pain, nausea, fatigue) as well as treatment's functional impact (eg ability to work, enjoy hobbies). Scale: 0-4. 0: Not at all, 4: Very much
  Values reported as "0.00 (0.00)" are accurate in all outcome measures.
Time Frame: Baseline, 3-month, 6-month, 12-month, 24-month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline; 3-month; 6-month; 12-month; 24-months: FACT-G (physical and functional well-being sections)
Arm/Group | Baseline | 3-month | 6-month | 12-month | 24-months
Number analyzed (Participants) | 9 | 8 | 7 | 6 | 1
score on a scale
  I have lack of energy | 0.67 (.47) | 1.63 (1.32) | 1.43 (0.90) | 1.67 (0.94) | 1.00 (0.00)
  I have nausea | 0.22 (0.42) | 0.38 (0.70) | 0.00 (0.00) | 0.50 (0.76) | 0.00 (0.00)
  Because of my physical condition, I have trouble meeting the needs of my family | 0.44 (0.83) | 1.00 (1.50) | 1.00 (1.41) | 0.67 (0.75) | 4.00 (0.00)
  I have pain | 0.33 (0.67) | 1.13 (1.17) | 1.43 (1.05) | 1.50 (0.50) | 4.00 (0.00)
  I am bothered by side effects of treatment | 0.22 (0.42) | 0.63 (0.70) | 0.71 (1.03) | 2.83 (0.69) | 0.00 (0.00)
  I feel ill | 0.11 (0.31) | 0.38 (0.70) | 0.14 (0.35) | 0.67 (1.49) | 0.00 (0.00)
  I am forced to spend time in bed | 0.22 (0.63) | 1.13 (1.54) | 0.57 (1.05) | 1.33 (1.60) | 3.00 (0.00)
  I am able to work (include work at home) | 3.00 (1.41) | 1.13 (1.54) | 2.57 (1.68) | 1.67 (1.70) | 0.00 (0.00)
  My work (include work at home) is fulfilling | 3.00 (1.33) | 2.88 (1.69) | 2.29 (1.58) | 1.83 (1.86) | 0.00 (0.00)
  I am able to enjoy life | 3.44 (0.96) | 3.38 (0.86) | 2.43 (1.18) | 2.17 (1.07) | 2.00 (0.00)
  I have accepted my illness | 3.00 (1.33) | 3.13 (1.27) | 2.71 (1.28) | 3.00 (1.00) | 3.00 (0.00)
  I am sleeping well | 3.33 (0.67) | 2.75 (0.97) | 1.71 (1.28) | 2.67 (1.25) | 1.00 (0.00)
  I am enjoying the things I usually do for fun | 3.33 (0.94) | 2.00 (1.66) | 2.29 (1.28) | 1.83 (1.21) | 0.00 (0.00)
  I am content with the quality of my life right now | 2.88 (1.69) | 2.00 (1.73) | 2.00 (1.60) | 2.17 (1.21) | 0.00 (0.00)

2. Primary Outcome: Assessment of Severity of Various Treatment-related Side Effects as Assessed by the FACT-En Questionnaire
Description: The Functional Assessment of Cancer Therapy - Endometrial (FACT-EN) questionnaire is a prospectively-validated questionnaire that asks patients to rated the severity of various possible treatment side effects (eg GI pain, pelvic pain, shortness of breath) Scale: 0-4. 0: Not at all, 4: Very much
Time Frame: Baseline, 3-month, 6-month, 12-month, 24-month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline; 3-month; 6-month; 12-month: FACT-En
- 24-months: FACT-G En
Arm/Group | Baseline | 3-month | 6-month | 12-month | 24-months
Number analyzed (Participants) | 9 | 8 | 7 | 6 | 1
score on a scale
  I have swelling in my stomach area | 0.44 (0.68) | 0.75 (1.09) | 0.43 (0.49) | 1.00 (1.15) | 0.00 (0.00)
  I have cramps in my stomach area | 0.11 (0.31) | 0.50 (0.71) | 0.14 (0.35) | 0.67 (1.11) | 0.00 (0.00)
  I have discomfort or pain in my stomach area | 0.33 (0.67) | 0.63 (0.86) | 0.43 (0.49) | 1.00 (1.15) | 0.00 (0.00)
  I have vaginal bleeding or spotting | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  I have vaginal discharge | 0.11 (0.31) | 0.13 (0.33) | 0.14 (0.35) | 0.00 (0.00) | 0.00 (0.00)
  I am unhappy about a change in my appearance | 0.22 (0.42) | 1.25 (1.64) | 0.71 (0.70) | 1.83 (1.67) | 0.00 (0.00)
  I have hot flashes/hot flushes | 0.56 (1.07) | 0.38 (0.48) | 0.43 (0.49) | 0.17 (0.37) | 0.00 (0.00)
  I have cold sweats | 0.11 (0.31) | 0.25 (0.43) | 0.00 (0.00) | 0.17 (0.37) | 0.00 (0.00)
  I have night sweats | 0.67 (1.05) | 0.75 (0.97) | 0.57 (0.73) | 0.50 (0.50) | 0.00 (0.00)
  I feel fatigued | 1.00 (0.94) | 1.25 (1.20) | 0.86 (0.83) | 1.67 (0.94) | 0.00 (0.00)
  I have pain or discomfort with intercourse | 0.11 (0.31) | 0.38 (0.99) | 0.14 (0.35) | 0.67 (1.49) | 0.00 (0.00)
  I have trouble digesting food | 0.00 (0.00) | 0.38 (0.70) | 0.29 (0.45) | 0.33 (0.47) | 0.00 (0.00)
  I have been short of breath | 0.33 (0.67) | 0.38 (0.48) | 0.14 (0.35) | 0.33 (0.47) | 0.00 (0.00)
  I am bothered by constipation | 1.22 (1.55) | 1.50 (1.73) | 0.43 (1.05) | 1.67 (1.70) | 3.00 (0.00)
  I urinate more frequently than usual | 0.56 (0.96) | 1.00 (1.00) | 0.86 (1.36) | 1.33 (1.11) | 0.00 (0.00)
  I have discomfort or pain in my pelvic area | 0.33 (0.67) | 1.13 (1.17) | 0.57 (1.05) | 0.67 (1.11) | 0.00 (0.00)

3. Primary Outcome: Assessment of Severity of Neurotoxicity Side Effects as Assessed by the FACT/GOG-NTX-4 Scale
Description: The Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity 4 Item Version (FACT/GOG-NTX-4) scale is a prospectively-validated questionnaire that assesses the severity of side effects related to neurotoxicity (paresthesia, pain in hands/feet) Scale: 0-4. 0: Not at all, 4: Very much
Time Frame: Baseline, 3-month, 6-month, 12-month, 24-month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline; 3-month; 6-month; 12-month; 24-months: FACT-GoG
Arm/Group | Baseline | 3-month | 6-month | 12-month | 24-months
Number analyzed (Participants) | 9 | 8 | 7 | 6 | 1
score on a scale
  I have numbness or tingling in my hands | 0.44 (0.68) | 1.63 (1.58) | 1.71 (1.28) | 2.33 (1.37) | 0.00 (0.00)
  I have numbness or tingling in my feet | 0.78 (1.03) | 2.50 (1.73) | 2.71 (1.03) | 3.17 (0.90) | 4.00 (0.00)
  I feel discomfort in my hands | 0.33 (0.67) | 0.88 (1.05) | 1.29 (0.88) | 1.67 (1.37) | 0.00 (0.00)
  I feel discomfort in my feet | 1.00 (1.25) | 1.88 (1.76) | 1.71 (1.48) | 2.83 (1.46) | 1.00 (0.00)

4. Primary Outcome: Assessment of Severity of GI Side Effects as Assessed by the FACT-C Questionnaire
Description: The Functional Assessment of Cancer Therapy - Colorectal (FACT-C) scale is a prospectively-validated questionnaire that asses GI-related side effects (diarrhea, fecal incontinence) Scale: 0-4. 0: Not at all, 4: Very much
Time Frame: Baseline, 3-month, 6-month, 12-month, 24-month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline; 3-month; 6-month; 12-month; 24-months: FACT-C (items C3 and C5)
Arm/Group | Baseline | 3-month | 6-month | 12-month | 24-months
Number analyzed (Participants) | 9 | 8 | 7 | 6 | 1
score on a scale
  I have control of my bowels | 4.00 (0.00) | 2.25 (1.79) | 2.57 (1.76) | 3.33 (0.94) | 4.00 (0.00)
  I have diarrhea | 0.56 (1.07) | 1.00 (1.50) | 0.43 (0.49) | 0.33 (0.47) | 0.00 (0.00)

ADVERSE EVENTS:
Time Frame: Baseline, 3-months, 6-months, 12-months, 24-months
Arm/Group | Quality of Life Evaluation
All-Cause Mortality (participants affected / at risk) | 1/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT04743999/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT04743999/ICF_002.pdf